CLINICAL TRIAL: NCT05207943
Title: Efficacy of the NXSignal Device for the Treatment of Anterior Cruciate Ligament Injuries. Randomized Controlled Clinical Trial
Brief Title: Efficacy of the NXSignal Device for the Treatment of Anterior Cruciate Ligament Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESALCA
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: physical therapy modality; Electric Stimulation Therapy; Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention to which the subjects have been assigned, the specialist and the researcher who collects the information and performs the follow-ups will be blinded, using the simulated NESA XSIGNAL® device. Data analysis will also be performed in a blinded fashion.
  Patients will be assigned to NESA XSIGNAL® device 1 or 2. These devices will be labeled "1" and "2" and only the manufacturer will know which is the real or the simulated one. In the same way, to avoid subjective comparisons of the participants, in the same room, device 1 and 2 at the same time will not be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-invasive Neuromodulation (Experimental): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level and and in the popliteal fossa.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Sham Comparator): Placebo microcurrents Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level and in the popliteal fossa.
  Interventions: Device: Placebo Non-invasive Neuromodulation
- Control (No Intervention): Participant will maintain the conventional rehabilitation treatment

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 10 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7. Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 millivolt and intensity 0.5 μA.
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but microcurrents device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
Injury to the anterior cruciate ligament (ACL) is very common among sports professionals and the general population [. Unlike other joint injuries, it is reversible, but it can damage adjacent tissues, particularly the meniscus, and catalyze knee osteoarthritis.

ACL injury produces instability, joint mechanical alteration, which can lead to degenerative joint diseases. The goal of treating the injury will be to prevent symptomatic instability, restore normal knee kinematics, and prevent degenerative joint disease .

Its usual treatment is surgical and therefore contributes to a significant cost for the health system, both for the surgeries themselves, and for the rehabilitation and subsequent recovery processes.

Within recovery therapies, in some cases, and given their popularity within the world of physiotherapy, electrotherapy techniques are proposed, primarily transcutaneous electrical nerve stimulation-type techniques with action on the muscular system and analgesia.

An early intervention with neuromuscular electrostimulation electrotherapy (NMES) combined with repeated exercises is effective for the recovery of strength and restoration of the biomechanical symmetry of the limb.

There is a diversity of opinions and disparate results regarding the use of this type of technique , in any case, it has been shown that electrical stimulation favors cell migration and joint tissue regeneration.

DETAILED DESCRIPTION:
The design of this study is a randomised, triple blind clinical trial with placebo control.

The general configuration of the study consists of capturing a group of patients treated with the same ACL surgical technique, operated on by the same surgeon, and including an additional treatment with the NESA XSIGNAL® device in a group of them.

For this, a double-blind capture system will be available (neither users nor specialists responsible for recovery will know which patients enter the complementary treatment) and two NESA XSIGNAL® devices operating double-blind (due to the imperceptivity of the stimulation performed, there will be a placebo machine and another that applies the treatment).

At the end of the study, the results obtained between the different groups of patients will be able to be compared; those additionally treated with a device, those treated with a placebo device and those in the standard rehabilitation procedure without a device.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years old
* In normal conditions and mentally competent to participate in the study.
* Not having previous knee surgeries.
* In condition to complete the study questionnaires.

Exclusion Criteria:

* Present some of the contraindications for a treatment with NESA XSIGNAL®: pacemakers, internal bleeding, do not apply electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and / or electricity phobia.
* Not having signed the informed consent.
* Urgent surgical interventions.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Knee circumference | Up to 4 month
  Centimeter measurement supra and infrapatellar with a tape measure with the leg in extension and without muscle contraction.
Motor Control | Up to 4 month
  It will be assessed through a dop jump, vertical jump test and Single leg squat.
Functional ability | Up to 4 month
  We will use the International Knee Documentation Committee (IKDC) questionnaire.
Level of Pain | Up to 4 month
  The Visual Analogue Scale (VAS) will be used to measure the perception of pain, which consists of a longitudinal line with 11 values ranging from 0 (none The Visual Analogue Scale (VAS) will be used to measure the perception of pain, which consists of a longitudinal line with 11 values ranging from 0 (no pain sensation) to 10 (maximum pain imaginable)

SECONDARY OUTCOMES:
Range of motion | Up to 4 month
  To measure this variable, we will use a goniometer, which will align its fixed arm with the proximal segment of the limb, and the mobile arm with the distal segment, making its axis coincide with the axis of knee movement . 3 measurements will be carried out actively and another 3 passively, choosing the highest value obtained for each one. Flexion and extension movements will be analyzed.
Brain activity | Up to 4 month
  Brain activity will be measured through an Electroencephalogram (EEG). Corresponds to a technique for studying the electrical activity of the brain through electrodes located on the scalp The parameters to be measured are the waves beta (13-30 Hz), which are produced when a subject is awake doing cognitive work and perceiving environmental stimulus
Quality of life related to health | Up to 4 month
  The SF-12 scale will be applied
Psychological perception test: | Up to 4 month
  TSK-11SV questionnaire (version adapted to Spanish). It is an 11-item questionnaire about fear of movement or injury. Patients have to indicate their degree of agreement with each of the statements presented, using a Likert-type scale from 1 (totally disagree) to 4 (totally agree). This questionnaire is designed to also assess the avoidance dimensions of activity and harm, but in this work we will only use the total score. High scores indicate greater fear of movement

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- University of Las Palmas de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Result] Stewart BA, Momaya AM, Silverstein MD, Lintner D. The Cost-Effectiveness of Anterior Cruciate Ligament Reconstruction in Competitive Athletes. Am J Sports Med. 2017 Jan;45(1):23-33. doi: 10.1177/0363546516664719. Epub 2016 Sep 30. PMID 27590175
- [Result] Kakavas G, Malliaropoulos N, Bikos G, Pruna R, Valle X, Tsaklis P, Maffulli N. Periodization in Anterior Cruciate Ligament Rehabilitation: A Novel Framework. Med Princ Pract. 2021;30(2):101-108. doi: 10.1159/000511228. Epub 2020 Dec 2. PMID 33264774
- [Result] van Melick N, van Cingel RE, Brooijmans F, Neeter C, van Tienen T, Hullegie W, Nijhuis-van der Sanden MW. Evidence-based clinical practice update: practice guidelines for anterior cruciate ligament rehabilitation based on a systematic review and multidisciplinary consensus. Br J Sports Med. 2016 Dec;50(24):1506-1515. doi: 10.1136/bjsports-2015-095898. Epub 2016 Aug 18. PMID 27539507